CLINICAL TRIAL: NCT04647994
Title: Exploratory Study in COVID-19 During Pregnancy
Brief Title: Exploratory Study: COVID-19 and Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 30270820.3.0000.0068
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Pregnant Women; Covid19
Keywords: pregnancy; SARS-CoV-2; vertical transmission
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Covid-19 HC patients: Pregnant women hospitalized with symptoms and diagnosis of SARS-CoV-2 at HC-FMUSP.
  Interventions: Diagnostic Test: SARS-CoV-2 serology
- Delivery patients: Asymptomatic pregnant women that tested SARS-CoV-2 serology (positive or negative serology) at the delivery time at Universitarian Hospital HU-USP and HC-FMUSP.
  Interventions: Diagnostic Test: SARS-CoV-2 serology
- Prenatal patients: Pregnant women that performs prenatal care in Universitarian Hospital HU-USP or HC-FMUSP with diagnosis of SARS-CoV-2.
  Interventions: Diagnostic Test: SARS-CoV-2 serology
- Negative serology patients: Pregnant women that performs prenatal care with symptoms and tested serology/swab negative for SARS-CoV-2.
  Interventions: Diagnostic Test: SARS-CoV-2 serology

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 serology — Serology test of SARS-CoV-2 for pregnant women

SUMMARY:
The SARS-CoV-2 infection may behave differently in pregnant and postpartum women in the short and long term. Several risk factors or medication use can interfere on disease' evolution and vertical transmission. Thus, due the current pandemic and the scarcity of scientific studies involving pregnant women with covid-19 or positive serology, combined with the need to elucidate the behavior of this viral infection in pregnant women in our population, this study aims to evaluate the clinical and laboratory evolution, transplacental passage, gestational and neonatal outcomes in pregnancies with positive SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with clinical symptoms or positive serology for SARS-CoV-2 hospitalized or in delivery time;
* Asymptomatic pregnant women for SARS-CoV-2 during pregnancy and hospitalized for delivery at HU-USP.
* Pregnant women diagnosed with SARS-CoV-2 prior to delivery and who, after the quarantine period, followed prenatal care and delivered at the HU-USP or HCFMUSP.

Exclusion Criteria:

* Non-confirmation of maternal SARS-CoV-2 infection in pregnant women hospitalized or in delivery time.
* Withdrawal of pregnant woman to continue in the study.

Ages: 17 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women with clinical symptoms or positive serology for SARS-CoV-2 hospitalized, in prenatal care, or in delivery time.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-11 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-13 (Estimated)

PRIMARY OUTCOMES:
Diagnostic test: SARS-CoV-2 serology | 01/07/2021
  Number of pregnant women with COVID-19 infection assessed with a serology test

SECONDARY OUTCOMES:
Laboratorial analysis of maternal and umbilical cord blood | 01/07/2021
  Number of participants with transplacental passage of SARS-CoV-2 assessed by laboratorial analysis of maternal and umbilical cord blood
Laboratorial analysis of Amniotic Fluid | 01/07/2021
  Number of participants with transplacental passage of SARS-CoV-2 assessed by amniotic fluid analysis
Placenta biopsy | 01/07/2021
  Number of participants with transplacental passage of SARS-CoV-2 assessed by placenta biopsy
Laboratorial analysis of colostrum | 01/07/2021
  Number of participants with transplacental passage of SARS-CoV-2 assessed by colostrum
Ovarian remains biopsy | 01/07/2021
  Number of participants with transplacental passage of SARS-CoV-2 assessed by ovarian remains biopsy in cases of abortion and fetal death.
Blood count analysis | 01/07/2021
  Number of participants with adverse events assessed by the blood count analysis after SARS-CoV-2 infection.
Laboratorial analysis of thyroid hormones | 01/07/2021
  Number of participants with adverse events assessed by the thyroid hormones analysis after SARS-CoV-2 infection.
PCR analysis | 01/07/2021
  Number of participants with adverse events assessed by the PCR analysis after SARS-CoV-2 infection.
Laboratorial analysis of Interleukins | 01/07/2021
  Number of participants with adverse events assessed by the interleukins analysis after SARS-CoV-2 infection.
Fetal morphology ultrasound | 01/07/2021
  Number of babies with developmental changes and fetal morphology alterations assessed by ultrasound after the maternal diagnosis of Covid-19.
Placental insufficiency ultrasound | 01/07/2021
  Number of participants with placental insufficiency and altered fetal well-being assessed by ultrasound after a positive maternal diagnosis of SARS-CoV-2.
Type of delivery | 01/07/2021
  Number of patients that performed natural delivery or caesarean, assessed by a structured questionnaire.
Gestational age at delivery | 01/07/2021
  Gestational age at delivery and premature cases, assessed by a structured questionnaire.
Apgar score | 01/07/2021
  Newborn's apgar score at first, second and third minutes after birth, assessed by a Apgar Score Scale (0 = minimum value and 10 = maximum value)
Newborn weight | 01/07/2021
  Newborn's weight immediately after birth, assessed by a pediatric weight balance
Fatigue Scale | 01/07/2021
  Number of patients with persistent symptoms of fatigue, assessed by a Fatigue Structured Scale
Prone Position | 01/07/2021
  Number of patients who needed intervention with a prone position during hospitalization, accessed by the medical record data.
Use of mechanical ventilation | 01/07/2021
  Number of patients who needed intervention with a mechanical ventilation and oxygen during hospitalization, accessed by the medical record data.
Pulmonary Ultrasound | 01/07/2021
  Number of patients with alterations in pulmonary ultrasound and chest tomography resulting from SARS-Cov2 infection.
Chest Tomography | 01/07/2021
  Number of patients with alterations in pulmonary ultrasound and chest tomography resulting from SARS-Cov2 infection.
Anxious and depressive symptoms - HAD questionnaire | 01/07/2021
  Number of patients with anxious and depressive symptoms in prenatal and postpartum, assessed by Hospital Anxiety and Depression Scale.
Heart rate variability electrocardiogram | 01/07/2021
  Number of patients with cardiac autonomic modulation, assessed by a heart rate variability electrocardiogram.
Laboratorial analysis of glycated hemoglobin | 01/07/2021
  Number of patients with endocrine system alterations after the Covid-19 infection, assessed by laboratorial analysis of glycated hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Rossana P Francisco, PhD, Principal Investigator — Faculdade de Medicina da Universidade de São Paulo - FMUSP
Locations (1):
- Rossana P Fracisco, São Paulo, Brazil